CLINICAL TRIAL: NCT03871634
Title: Assessment of Nutritional Status of Patients With Crohn's Disease
Status: Completed | Type: Observational
Sponsor: Harokopio University (Other)
Collaborators: Evangelismos Hospital (Other); Sotiria General Hospital (Other); General Hospital of Nikaia "Saint Panteleimon" (Other)
Responsible Party: Principal Investigator, Meropi Kontogianni, Associate Professor of Clinical Nutrition, Harokopio University
Other Study IDs: 122
Record Dates: First submitted 2019-03-09; First posted 2019-03-12 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Crohn's Disease; Malnutrition; Overweight and Obesity; Sarcopenia; Sarcopenic Obesity
MeSH Terms: conditions — Crohn Disease; Malnutrition; Overweight; Obesity; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Good nutritional status of patients with Crohn's disease (CD) is associated with better outcome of the disease and better health-related quality of life. The prevalence of malnutrition in patients with Crohn's disease varies and is higher in patients with active disease. Available studies in the literature have assessed the nutritional status of patients with Crohn's disease. However, sample size of available studies is small and highly heterogeneous, and most patients are hospitalized with active disease. The aim of the present study is a thorough assessment of nutritional status of 250 patients either with active Crohn's disease or in remission of the disease using multiple widely available tools and methods, in order to assess their accuracy and estimate the prevalence of multiple malnutrition phenotypes such as undernutrition, sarcopenia, sarcopenic obesity and cachexia as well as overweight and obesity. Finally, the effect of the nutritional status on the course of the disease will be investigated.

DETAILED DESCRIPTION:
The study sample will comprise of 250 adults with proven Crohn's disease, either with active disease or in remission phase. A detailed medical and nutritional assessment will be implemented at baseline. Data regarding the hospitalizations, disease relapse, duration of remission and complications of all the patients will be collected one year after the baseline assessment.

More specifically regarding the detailed assessment, firstly, gastroenterologists of the research team will complete a full medical record regarding the localization of the disease, activity of disease (active or remission), complications, comorbidities and medication. The activity of Crohn's disease will be assessed using the Harvey-Bradshaw Index (HBI). Blood will be collected for all patients with Crohn's Disease.

Furthermore, in the Laboratory of Clinical Nutrition & Dietetics at Harokopio University, patients will participate in the following procedures:

* Indirect calorimetry: Resting Energy Expenditure (REE) measurement will be performed (Ultima Series, MedGraphics Cardiorespiratory Diagnostics).
* Anthropometry: Weight, height, waist and mid-arm circumference, and triceps skinfold will be measured. Body mass index, mid-arm muscle circumference and area will be estimated using standard equations.
* Body composition analysis and bone density measurement: Total body Dual-energy X-Ray Absorptiometry (DXA) and Spine (Lunar DPX-MD, Madison, WI, USA) will be performed.
* Muscle strength and performance status: Handgrip strength measurement based on certain protocol and the "Short Physical Performance Battery" (SPPB) tool will be implemented.
* Dietary intake evaluation: A Food-Frequency Questionnaire (FFQ) and two non-consecutive 24h recalls (one weekday and one weekend day) will be recorded. Data will be analyzed to estimate energy, macro- and micronutrients intake (Nutritionist Pro software, 2.2 version). Food group intake, meal patterns and MedDietScore will also be evaluated.
* Physical activity assessment: Patients' physical activity levels will be assessed using the "Harokopio Physical Activity Questionnaire".
* Fatigue and Quality of Life Assessment: Assessment of fatigue will be performed with "Fatigue Severity Scale" (FSS), when assessment of quality of life with be performed with "Food Related Quality of Life" (FR-QoL) and "Short Inflammatory Bowel Disease Questionnaire" (SIBDQ).

In addition, patients' nutritional risk or nutritional status will be assessed through several previously validated tools like the Subjective Global Assessment, the Nutrition Risk Score 2002, the Malnutrition Universal Screening Tool, the efficacy of which will be tested in the present study. Patients will be also categorized according to GLIM criteria for the diagnosis of malnutrition.

Six months and twelve months after the baseline assessment of the study samples, data will be collected regarding the hospitalizations, disease relapse, duration of remission and complications of all the patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults with Crohn's Disease either with active disease or in remission phase.

Exclusion Criteria:

* Hospitalized patients
* Patients with Crohn's disease <6 months
* Patients with cancer
* Patients with heart insufficiency
* Patients with renal insufficiency
* Patients with short bowel syndrome (SBS)
* Patients with parenteral nutrition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 250 adult patients with active Crohn's Disease or in remission phase
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of malnutrition phenotypes | Baseline
  Prevalence of different malnutrition phenotypes (e.g. undernutrition, sarcopenia, sarcopenic obesity), in crohn disease patients either with active disease or in remission, by implementing a thorough nutritional assessment.

SECONDARY OUTCOMES:
Validity test of available tools | Baseline
  Test the sensitivity, specificity, positive and negative prognostic values of already available tools for nutritional screening or assessment against a combined index as the reference tool. If no tool is estimated as valid, a new combination of nutritional, biochemical and/or clinical parameters will be synthesized and its validity as a new screening or assessment tool will be assessed for the detection of cirrhotic patients at risk of malnutrition or already malnourished.

CONTACTS AND LOCATIONS:
Locations (1):
- Harokopio University, Athens, Kallithea, Greece